CLINICAL TRIAL: NCT01183065
Title: A Multi-Institution Phase II Study of Pralatrexate With Vitamin B12 and Folic Acid Supplementation for Previously Treated Recurrent or Metastatic Head and Neck Squamous Cell Cancer (HNSCC)
Brief Title: Study of Pralatrexate With Vitamin B12 and Folic Acid Supplementation for Previously Treated Recurrent or Metastatic Head and Neck Squamous Cell Cancer (HNSCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York University Cancer Institute (Other); NYU Langone Health (Other); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-112
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Head and Neck Cancer
Keywords: Pralatrexate; Vitamin B12; Folic Acid; 10-112
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid; Therapeutics

ARMS (1):
- pralatrexate and vitamin supplementation (Experimental): This will be an open-label, single arm, Simon optimal two-stage design phase II study.
  Interventions: Drug: Pralatrexate With Vitamin B12 and Folic Acid

INTERVENTIONS:
Drug: Pralatrexate With Vitamin B12 and Folic Acid — Patients will be treated with 30 mg/m2 of pralatrexate intravenously once weekly for 3 weeks in a 4 week cycle with vitamin supplementation. Patients will take 1.0-1.25 mg oral folic acid on a daily basis. Folic acid should be initiated during the 10-day period preceding the first dose of pralatrexate and dosing will be continued during the full course of therapy and for 30 days after the last dose of pralatrexate. Patients will also receive a vitamin B12 (1 mg) intramuscular injection no more than 10 weeks prior to the first dose of pralatrexate and every 8-10 weeks thereafter. Subsequent vitamin B12 injections may be given the same day as treatment with pralatrexate.
  Other Names: Radiologic assessment of disease will be conducted every 1.5 to 2 cycles (approximately; every 6 to 8 weeks); after 6 months, radiologic studies will be performed every 2.5 to 3; cycles (approximately every 10 to 12 weeks) of therapy.

SUMMARY:
The purpose of this study is to find out if the experimental drug pralatrexate with the vitamins folic acid and vitamin B12 might be an effective treatment for head and neck cancer. The reason we are doing this study is because another drug called methotrexate has been used for a long time to treat head and neck cancer patients. Pralatrexate was designed by scientists to be a new drug that works better than methotrexate. Laboratory studies have shown that pralatrexate works better than methotrexate at killing cancer cells.

Pralatrexate has already been studied in patients with other types of cancers, such as lymphoma and lung cancer. The results from those studies were promising. Pralatrexate was recently approved by the Food and Drug Administration (FDA) as a new treatment for a cancer called peripheral T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically confirmed recurrent and/or metastatic squamous cell carcinoma of the head and neck, including unknown primary squamous cell carcinomas of the neck. Confirmation of biopsy/diagnosis will be performed at MSKCC or at participating sites (NYU Cancer Institute/NYU Medical Center/ Bellevue Hospital Center).
* Patients must be at least 18 years of age.
* ECOG performance status must be ≥ 0 or 1.
* Disease must be measurable by RECIST version 1.1 criteria.
* Patients must have been previously treated with systemic chemotherapy (i.e., chemotherapy and/or targeted therapies such as cetuximab for recurrent/metastatic HNSCC,.
* At least four weeks must have elapsed from previous radiation therapy. Patients must have recovered from the acute toxic effects of treatment prior to study enrollment.
* Patients must have adequate organ function, as follows:

Adequate bone marrow reserve: absolute neutrophil count (ANC) > 1,000 cells/mm3, platelets > 100,000 cells/mm3, and hemoglobin > 9 g/dL Hepatic: AST and ALT ≤ 3 X upper limit of normal (ULN); AST and ALT ≤ 5 X ULN if liver metastasis present; Total bilirubin ≤ 1.5 x ULN unless Gilbert's disease is present Renal: Serum creatinine ≤ 1.5 mg/dL or creatinine clearance (by either 24 hour urine collection or Cockcroft-Gault equation) > or = to 55 ml/min

* Both women and men and members of all races and ethnic groups are eligible for this trial.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Both men and women must agree to use a reliable method of birth control until 30 days following the last dose of study drug.

Exclusion Criteria:

* History of any brain metastases unless resected with no evidence for > 12 weeks and not on steroids
* Women who are lactating
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment and safety analysis
* Patients who have undergone an allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pralatrexate and Vitamin Supplementation
Started | 13
Completed | 12
Not Completed | 1
Not completed — Patient no longer fits eligibility crite | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pralatrexate and Vitamin Supplementation
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Overall Response Rate (CR+PR)
Description: by RECIST version 1.1 criteria
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Pralatrexate and Vitamin Supplementation
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Arm/Group | Pralatrexate and Vitamin Supplementation
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate and Vitamin Supplementation (N=12)
Injury/poison & proced complications Other, spec (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate and Vitamin Supplementation (N=12)
Alkaline phosphatase increased (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (5)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes